CLINICAL TRIAL: NCT05621798
Title: Quantifying the Benefits and Cost-effectiveness of Real-Ear Measurements (REM) for Hearing Aid Fitting
Acronym: BREM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5551888
Record Dates: First submitted 2022-08-11; First posted 2022-11-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: REM; Real Ear Measurements; Sensorineural Hearing Loss; Hearing Aid Fitting; Speech Intelligibility Tests in Noise; HERE; SSQ-49
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Sleep, REM

STUDY DESIGN:
Intervention Model Description: On the first fit visit the participants will be fitted either with the manufacturers "first-fit" or "initial fit" program or using the REM measurements. We will randomize all patients into two groups; Half of the participants will be fitted with the Phonak "first fit" fitting rule and the other half using the Phonak TargetMatch that utilizes REM fitting. After around 2-3 months, depending on the clinic schedule, the participants will be crossed-over to the other method, so that the group that first got the manufacturers fit will now receive the fit based on REM and vice versa. Third visit will take place 2-3 months after the second visit and the participants will get to choose which fit they will prefer for their hearing aids. Fourth visit takes place around 6 months after the third visit when the participants have been wearing their hearing aids for a year.
Who Masked: Participant, Care Provider
Masking Description: Patients are having their hearing aids fitted by manufacturer's initial fit method or by REM. In both fittings participants will be hearing sounds at different intensities and frequencies but they are unaware of the exact fitting method used. The "first fit" and REM measurement sounds and procedures are different, but for first-time users unknown. Both procedures are conducted by audiologist but only the other of the fitting results is being used for the hearing aid adjusting. During the next fitting appointment the participant is also seen and the hearing aid is re-fitted by another audiologist than the first time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hearing Aid Manufacturer's Software Group (Active Comparator): Participants' hearing aids are fitted by using manufacturer's software.
  Interventions: Other: Hearing Aid Manufacturer's Software; Other: REM (Real Ear Measurements)
- REM Group (Active Comparator): Participants' hearing aids are fitted by REM (Real Ear Measurements) method.
  Interventions: Other: Hearing Aid Manufacturer's Software; Other: REM (Real Ear Measurements)

INTERVENTIONS:
Other: Hearing Aid Manufacturer's Software — When using hearing aid manufacturer's software (s.c. "first-fit" or "initial fit") the fitting will follow the guided fitting procedure in the fitting software.
Other: REM (Real Ear Measurements) — Participants' hearing aids are fitted by using REM. In this method REM measurement tube is placed inside participant's ear canal near the tympanic membrane and the Real Ear Unaided Gain (REUG) is measured. REUG is used to measure the ear canal without any hearing device and shows the patients ear acoustics. Next the hearing aid is placed on the patients ear together with the REM measurement tube. In REM measurements the Real-Ear Occluded Gain (REOG) is measured with the hearing aid off. REOG allows consideration of the attenuation caused by the earpiece and its obstructing effect of external sounds. Next Real Ear Aided Response (REAR) is measured with the hearing device on. REAR allows measurement of the hearing device's amplification effect within the patients' ear and includes the effect of the patient's ear acoustics.

SUMMARY:
Adjusting hearing aid user's real ear performance by using probe-microphone technology (real ear measurement, REM) has been a well-known procedure that verifies whether the output of the hearing aid at the eardrum matches the desired prescribed target. Still less than half of audiologists verify hearing aid fitting to match the prescribed target amplification with this technology. Recent studies have demonstrated failures to match the prescribed amplification targets, using exclusively the predictions of the proprietary software. American Speech-Language-Hearing Association (ASHA) and American Academy of Audiology (AAA) have created Best Practice Guidelines that recommend using real-ear measurement (REM) over initial fit approach and also the recent ISO 21388:2020 on hearing aid fitting management recommends the routine use of REM. Still audiologists prefer to rely on the manufacturer's default "first-fit" settings because of the lack of proof over cost-effectiveness and patient outcome in using REM. There are only few publications of varying levels of evidence indicating benefits of REM-fitted hearing aids with respect to patient outcomes that include self-reported listening ability, speech intelligibility in quiet and noise and patients' preference. Our main research question is whether REM-based fitting improves the patient reported outcome measures - PROMs (SSQ, HERE) and performance-based outcome measures (speech-reception threshold in noise) over initial fit approach. An additional research question is whether REM-based fitting improves hearing aid usage (self-reported & log-data report). Eventually, the investigators will calculate the cost-effectiveness of REM-based fitting.

DETAILED DESCRIPTION:
Adjusting hearing aid user's real ear performance by using probe-microphone technology (real ear measurement, REM) has been a well-known procedure over 30 years among audiologists. With this measurement technique, it is possible to verify whether the output of the hearing aid at the eardrum matches the desired prescribed target. Still less than half of audiologists verify their hearing aid fitting to match the prescribed target amplification with this technology. Many still rely on the manufacturer's default "first-fit" settings (initial fit approach) which means that the patient's hearing thresholds at any given frequency are transferred to the programming software that predicts the output and gain of the hearing aid by using proprietary or modified prescriptive algorithm. These proprietary algorithms create an approximation over patients in situ hearing aid gain and output based on data such as the age of the patient, an estimate of microphone location effects, the ear mold or shell design and length, venting size, and tubing characteristics.

Recent studies have demonstrated failures to match the prescribed amplification targets, using exclusively the predictions of the proprietary software. The American Speech-Language-Hearing Association (ASHA) and American Academy of Audiology (AAA) have created Best Practice Guidelines that recommend using real-ear measurement (REM) over initial fit approach in order to verify the prescribed gain and output of the hearing aids. Accordingly, the recent ISO 21388:2020 on hearing aid fitting management recommends the routine use of REM. So why is REM still rarely applied clinically? The main reason is the lack of proof over cost-effectiveness and patient outcome. There are only few publications of varying levels of evidence indicating benefits of REM-fitted hearing aids with respect to patient outcomes that include self-reported listening ability, speech intelligibility in quiet and noise and patients' preference. According to a very recent systematic review and meta-analyses by Almufarrij et al. published in 2021, there are only six publications that meets the inclusion criteria, and the evidence favors REM fitting for all outcomes reported (self-reported listening ability, speech intelligibility in quiet and noise and preference). Still, the quality of evidence varies across the outcomes since all articles had a rather limited number of participants and only two used power calculation to determine the sample size. None of these studies reported health-related quality of life, which was assessed to be the primary outcome by the reviewers. Also, secondary outcomes of interest including adverse events, generic quality of life and cost-effectiveness were not assessed. The authors also acknowledged the lack of sufficient follow-up duration (the maximum duration was only 6 weeks) and the lack of permission for further adjustment to the amplification characteristics. In addition, the included studies failed to investigate first-time users over experienced hearing-aid users and the amplification characteristics the experienced users were familiar with, were not reported. This was judged to possibly impact on short-term outcomes since changes of hearing-aid users' amplification characteristics that they are already accustomed to, can cause discomfort. The authors also claimed that future studies should also estimate the importance of any benefit found and evaluate the reasons why participants are reporting these benefits.

In summary, current evidence indicates that the initial fit approach often fails to achieve the prescriptive acoustic gain and output of hearing aids, however, evidence which would clearly show that REM-based hearing aid fitting (which is time-consuming) is clinically relevant and cost-effective is lacking, and thus warrants further studies.

Our main research question is whether REM-based fitting improves the patient reported outcome measures - PROMs (SSQ, HERE) and performance-based outcome measures (speech-reception threshold in noise) over initial fit approach. These are the primary outcomes of our study. An additional research question is whether REM-based fitting improves hearing aid usage (self-reported & log-data report). Eventually, the investigators will calculate the cost-effectiveness of REM-based fitting. These are the secondary outcomes of our study.

ELIGIBILITY:
Inclusion Criteria:

* all first-time adult patients (18-80 years of age) eligible for bilateral hearing aid rehabilitation based on an evaluation by an otolaryngologist or an audiologist

Exclusion Criteria:

* confirmed cases of cognitive decline or dementia
* unilateral or conductive hearing impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Related Outcome Measure: Speech, Spatial and Qualities of Hearing Scale (SSQ) | Change measures: 0 months, 2 months, 4 months, 6 months.
  Participants are asked to fill out SSQ questionnaire during every clinical visit. This questionnaire includes 49 items with a numeric rating scale from 0 to 10 for each item and allows the assessment of hearing with and without hearing aids. Higher scores mean better outcome.
Patient Related Outcome Measure: Hearing in Real-Life Environments (HERE) | Change measures: 0 months, 2 months, 4 months, 6 months.
  Participants are asked to fill out HERE questionnaire during every clinical visit. Questionnaire includes 15 items with a numeric rating scale from 0 to 10 for each item and allows the assessment of hearing with and without hearing aids. Higher scores mean worse outcome.
Performance-based Outcome: Finnish matrix Sentence Test (FMST) | Change measures: 0 months, 2 months, 4 months, 6 months.
  Participants will conduct Finnish Matrix Sentence Test (FMST) during every clinical visit. This test measures participants' speech perception in noise.
Performance-based Outcome: Digit Triple Test (DTT) | Change measures: 0 months, 2 months, 4 months, 6 months.
  Participants will conduct Digit Triple Test (DTT) during every clinical visit. This test measures participants' speech perception in noise.

SECONDARY OUTCOMES:
Objective differences of the fitting parameters | Change measures: 0 months and 2 months
  Difference in desibel levels between initial fit and REM
Fitting preference | 12 months after the beginning of clinical visits
  Participants' preferences are measured by likert scale (1-10).
Hearing aid usage | 12 months after the beginning of clinical visits
  Participants' self-reported hearing aid usage and log-data report are recorded.
Cost effectiveness | Between 0-12 months.
  Additional time consumption for REM and number of additional contacts to the clinic are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aarno Dietz, Prof., Study Chair — ENT specialist; Matti Iso-Mustajärvi, Ass. prof., Study Director — ENT specialist; Laura Ihalainen, MD, Principal Investigator — ENT specialist; Tytti Willberg, PhD, Study Director — ENT specialist; Pia Linder, PhD, Study Director — Medical engineer
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams HB, Chisolm TH, McManus M, McArdle R. Initial-fit approach versus verified prescription: comparing self-perceived hearing aid benefit. J Am Acad Audiol. 2012 Nov-Dec;23(10):768-78. doi: 10.3766/jaaa.23.10.3. PMID 23169194
- [Background] Almufarrij I, Dillon H, Munro KJ. Does Probe-Tube Verification of Real-Ear Hearing Aid Amplification Characteristics Improve Outcomes in Adults? A Systematic Review and Meta-Analysis. Trends Hear. 2021 Jan-Dec;25:2331216521999563. doi: 10.1177/2331216521999563. PMID 33899603
- [Background] Almufarrij I, Munro KJ, Dillon H. Does probe-tube verification of real-ear hearing aid amplification characteristics improve outcomes in adult hearing aid users? A protocol for a systematic review. BMJ Open. 2020 Jul 19;10(7):e038113. doi: 10.1136/bmjopen-2020-038113. PMID 32690533
- [Background] Denys S, Latzel M, Francart T, Wouters J. A preliminary investigation into hearing aid fitting based on automated real-ear measurements integrated in the fitting software: test-retest reliability, matching accuracy and perceptual outcomes. Int J Audiol. 2019 Mar;58(3):132-140. doi: 10.1080/14992027.2018.1543958. Epub 2018 Dec 4. PMID 30513024
- [Background] Scollie S, Ching TY, Seewald R, Dillon H, Britton L, Steinberg J, Corcoran J. Evaluation of the NAL-NL1 and DSL v4.1 prescriptions for children: Preference in real world use. Int J Audiol. 2010 Jan;49 Suppl 1:S49-63. doi: 10.3109/14992020903148038. PMID 20109089
- [Background] Hawkings DP, Cook JA. Hearing aid software predictive gain values: How accurate are they? The Hearing Journal. 2003; 56(7): 26-34.
- [Background] Aarts NL, Caffee CS. Manufacturer predicted and measured REAR values in adult hearing aid fitting: accuracy and clinical usefulness. Int J Audiol. 2005 May;44(5):293-301. doi: 10.1080/14992020500057830. PMID 16028792
- [Background] Aazh H, Moore BC, Prasher D. Real ear measurement methods for open fit hearing aids: modified pressure concurrent equalization (MPCE) versus modified pressure stored equalization (MPSE). Int J Audiol. 2012 Feb;51(2):103-7. doi: 10.3109/14992027.2011.609182. Epub 2011 Oct 24. PMID 22023487
- [Background] Aazh H, Moore BC. The value of routine real ear measurement of the gain of digital hearing aids. J Am Acad Audiol. 2007 Sep;18(8):653-64. doi: 10.3766/jaaa.18.8.3. PMID 18326152
- [Background] Mueller HG, Picou EM. Survey examines popularity of real-ear probe-microphone measures. Hearing Journal. 2010; 63(5): 27-32.
- [Background] Valente M, Oeding K, Brockmeyer A, Smith S, Kallogjeri D. Differences in Word and Phoneme Recognition in Quiet, Sentence Recognition in Noise, and Subjective Outcomes between Manufacturer First-Fit and Hearing Aids Programmed to NAL-NL2 Using Real-Ear Measures. J Am Acad Audiol. 2018 Sep;29(8):706-721. doi: 10.3766/jaaa.17005. PMID 30222541
- [Background] Walravens E, Keidser G, Hickson L. Consistency of Hearing Aid Setting Preference in Simulated Real-World Environments: Implications for Trainable Hearing Aids. Trends Hear. 2020 Jan-Dec;24:2331216520933392. doi: 10.1177/2331216520933392. PMID 32602407